CLINICAL TRIAL: NCT04132167
Title: Supervised Perturbation Training Results in Changes in Balance and Falling in Patients With Multiple Sclerosis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Suleyman Demirel University (Other)
Responsible Party: Principal Investigator, HATİCE YAKUT, Principal investigator, Suleyman Demirel University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 12345
Record Dates: First submitted 2017-11-23; First posted 2019-10-18 (Actual); Last update posted 2019-10-25 (Actual); Status verified 2019-10

CONDITIONS: Multiple Sclerosis
Keywords: Rehabilitation; Multiple sclerosis; Tailored interventions
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- training group (Experimental): perturbation balance training
  Interventions: Procedure: perturbation training
- control group (Active Comparator): traditional physical therapy that including strengthening and stretching
  Interventions: Procedure: perturbation training

INTERVENTIONS:
Procedure: perturbation training — exercises for body stability in different positions (bridge, sitting, quadrupedal, half- kneeling, kneeling, standing, monopodalic) performed with visual biofeedback; transfers training performed in front of a mirror; ambulation training with courses drawn on the ground in a straight line and with more complex tracks with visual controlin particular using the protocols seated balance/strength training, standing bal- ance/weight-bearing training, mobility training and closed-chain training;

SUMMARY:
Physical exercise can prevent falls, certain types of exercise may be more effective. Perturbation-based balance training is a novel intervention involving repeated postural perturbations aiming to improve control of rapid balance reactions. The purpose of this study was to estimate the effect of perturbation- based balance training on falls and balance in daily life.Thirty patients with multiple sclerosis (PwMS) will assess with regard to dynamic balance, walking and falling. Patients randomly will allocate to a personalized (PRG) or traditional (TRG) rehabilitation group.

DETAILED DESCRIPTION:
Thirty patients with multiple sclerosis (PwMS) will assess with regard to dynamic balance, walking and falling. Patients randomly will allocate to a personalized (PRG) or traditional (TRG) rehabilitation group.

ELIGIBILITY:
Inclusion Criteria:

* An age older than 18 years
* Stable phase of the disease without relapses or worsening in the last three months
* Referring fear of falling or a history of falls (at least one fall in the last year).
* Individuals with a high level of balance.

Exclusion Criteria:

* Psychiatric disorders
* Blurred vision
* Severe cognitive impairment
* Severely impaired upright postural control or limited participation in a rehabilitation program
* Cardiovascular and respiratory disorders.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 15 (Estimated)
Dates: Start 2018-11-20 (Actual); Primary Completion 2019-10-20 (Estimated); Study Completion 2019-12-20 (Estimated)

PRIMARY OUTCOMES:
dynamic balance | 6 week
  the effects of perturbation dynamic balance training assessed with four square step test >15 seconds = increased risk of falls
walking | 6 week
  the effects of perturbation dynamic balance training assessed with 10 meter walking test
walking | 6 week
  the effects of perturbation dynamic balance training assessed with time up and go test(TUG).A score of 30 seconds or more suggests that the person may be prone to falls
falling | 6 week
  the effects of perturbation dynamic balance training assessed with Falling Efficacy Scale(FES). The FES is a 10-item test. On a scale from 1 to 10, with 1 being very confident and 10 being not confident at all.
fear of falling | 6 week
  The short FES-I is a 7-item self-report questionnaire for measuring perceived self-efficacy to avoid a fall in various situations

CONTACTS AND LOCATIONS:
Locations (1):
- Hatice Yakut, Isparta, Turkey (Türkiye)